CLINICAL TRIAL: NCT04668937
Title: Conséquences of the COVID-19 Lockdown Measures on the CHRU Nancy
Brief Title: Conséquences of the COVID-19 Lockdown Measures on the CHRU Nancy Pediatric Emergency Services
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BELIN Delphine, clinician, Central Hospital, Nancy, France
Other Study IDs: 2020PI235
Record Dates: First submitted 2020-12-11; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Number of Patients During the Studying Period; Reason for Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children who came to the Nancy's Pediatric emergencies during the study period in 2019
- Children who came to the Nancy's Pediatric emergencies during the study period in 2020

SUMMARY:
The first period of COVID 19 Lockdown Measures (From 18 March to 11 may 2020) change the French people way of life and their medicine knowledges. A study which evaluates the Nancy's Pediatric emergencies population utilization during this time could detect pathological changes. The medical impact of Home Confinement will show an increase (trauma, maltreatment) or decrease (virus disease) of several pathology. The study aims to help clinicians to the children care if another time of Home Confinement happened. The main objective is to evaluate the behavioural changes and the reason consultation in Nancy's Pediatric Emergencies from 18 March to 30 June 2020 comparate to the same time in 2019. We will continue the search after the end of Home Confinement until 30 June 2020 to evaluate what happened just after.

ELIGIBILITY:
Inclusion Criteria:

* children who are cared during the study period to the Nancy's pediatric emergencies

Exclusion Criteria:

* be more than 18 years old
* Not being seen by a doctor

Max Age: 17 Years | Sex: All
Age Groups: Child
Study Population: All children who came to the Nancy's Pediatric emergencies during the period of the 18 march to the 30 June 2019 and 2020
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patient who came to Nancy's pediatric emergencies during the study period | from 18 March to 30 June 2019 and 2020
Reason of consultation during the study period | from 18 March to 30 June 2019 and 2020

SECONDARY OUTCOMES:
Number of children who was send by a General practician | from 18 March to 30 June 2019 and 2020
Medical reason to be sending by a General practician | from 18 March to 30 June 2019 and 2020

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy's Pediatric Emergencies, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided